CLINICAL TRIAL: NCT04693663
Title: Treatment of Residual Myopic Refraction After 6 Months on Pseudophakic Patients Using Relex-Smile
Acronym: Relex-Smile
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Eye Hospital Pristina Kosovo (Other)
Responsible Party: Principal Investigator, Dr. Faruk Semiz, Head of Ophthalmology Department, Eye Hospital Pristina Kosovo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EHP
Record Dates: First submitted 2020-12-25; First posted 2021-01-05 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Pseudophakia; Myopia
MeSH Terms: conditions — Pseudophakia; Myopia

STUDY DESIGN:
Intervention Model Description: One group consisting of 40 eyes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ReLex Smile surgery (Other): Procedure/Surgery: Relex Smile The residual myopic refraction on Pseudophakic patients after 6 months using Relex-Smile surgery by VisuMax femtosecond laser. The residual refractive power was between -0.75D till -5.50D.The optical zone (lenticule diameter) and cap diameter were 6.5 and 7.5 mm respectively. After dissection of both anterior and posterior planes, the lenticule was extracted through 120 degree superior 3.5 mm incision and marked with a sterile marker(Viscot-Medster).
  Interventions: Procedure: Relex-Smile surgery

INTERVENTIONS:
Procedure: Relex-Smile surgery — surgery using Relex-Smile
  Other Names: Relex smile surgery

SUMMARY:
The aim of this study is to assess visual and refractive outcomes after laser vision correction (LVC) - ReLex Smile to correct residual myopic refraction after 6 months of pseudophakic (IOL) implantation.

Before SMILE YAG-Laser capsulotomy should be performed on all patients, regardless of posterior capsule ossification, in pseudophakic patients with residual refraction. When the YAG Laser is applied after the SMILE, there will be a diopter change.

DETAILED DESCRIPTION:
The residual myopic refraction after 6 month on pseudophakic patients using Relex-Smile surgery using VisuMax Femtosecond Laser.The residual myopic refractive power is between -0.75D till -5.50D.The optical zone(lenticule diameter) and cap diameter were 6.5 and 7.5 mm respectively.After dissection of both anterior and posterior planes, the lenticule was extracted through 120 degree superior 3.5mm incision and marked with a sterile marker(Viscot-Medster)

ELIGIBILITY:
Inclusion Criteria:

* residual myopic refraction -0.75d till -5.50D
* complain visual acuity regarding residual myopic refraction

Exclusion Criteria:

* active anterior segment pathologic features
* previous corneal or anterior segment surgery
* glaucoma
* history of ocular inflammation

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Increase of visual acuity | 6 months
  Treatment of residual myopic refraction on Pseudophakic patients, was performed using ReLex Smile after 6 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Eye Hospital Pristina, Pristina, Kosovo

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Semiz F, Lokaj AS, Musa NH, Semiz CE, Demirsoy ZA, Semiz O. SMILE for the Treatment of Residual Refractive Error After Cataract Surgery. Ophthalmol Ther. 2022 Aug;11(4):1539-1550. doi: 10.1007/s40123-022-00526-7. Epub 2022 May 28. PMID 35643966